CLINICAL TRIAL: NCT02438709
Title: Application of COX-2 Inhibitor for Treatment of Primary Hypertrophic Osteoarthropathy
Brief Title: Effect Observation Study of COX-2 Inhibitor to Treat Primary Hypertrophic Osteoarthropathy
Acronym: EOSCITPHO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 81170805，2008ZX09312-016
Record Dates: First submitted 2015-01-08; First posted 2015-05-08 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-04

CONDITIONS: Primary Hypertrophic Osteoarthropathy
MeSH Terms: conditions — Osteoarthropathy, Primary Hypertrophic | interventions — Cyclooxygenase 2 Inhibitors; Etoricoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- COX-2 Inhibitor (Experimental): Patients who take COX-2 inhibitor
  Interventions: Drug: COX-2 inhibitor

INTERVENTIONS:
Drug: COX-2 inhibitor — oral COX-2 inhibitor intake 60mg qd
  Other Names: EtoriCoxib

SUMMARY:
The purpose of this study is to determine whether COX-2 inhibitor is effective in the treatment of primary hypertrophic osteoarthropathy

DETAILED DESCRIPTION:
Patients with primary hypertrophic osteoarthropathy(PHO) were diagnosed based on clinical manifestations and symptoms. PHO patients were treated with COX-2 inhibitor after signing informed consent. The extend of alleviation, the change of the markers on prostaglandin E metabolic pathway and the adverse event on different time points were recorded to identify the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with primary hypertrophic osteoarthropathy clinically
* over 16 years old
* no other medication intake
* informed consent signed

Exclusion Criteria:

* below 16 years old
* active gastric ulcer
* inflammatory bowel disease
* New York Heart Association classification（NYHA） II to IV
* liver or renal failure
* allergic to nonsteroid anti-inflammatory drugs
* not willing to participate

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-12; Primary Completion 2015-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Prostaglandin E2（PGE2） level change after COX-2 inhibitor treatment in PHO patients | 3 months
  measure the serum prostaglandin E2 level at 3 months
Prostaglandin E2（PGE2） level change after COX-2 inhibitor treatment in PHO | 6 months
  measure the serum prostaglandin E2 level at 6 months

SECONDARY OUTCOMES:
change in pain on VAS scale after COX-2 inhibitor treatment | 3 months
  use Visual Analogue Score (VAS) to evaluate pain
change in pain on VAS scale after COX-2 inhibitor treatment | 6 months
change in pain on VAS scale after COX-2 inhibitor treatment | 12 months
The volume of distal part of middle finger change after COX-2 inhibitor treatment | 3 months
  Both left and right fingers were measured twice and the average value was defined as volume of distal part of middle finger
The volume of distal part of middle finger change after COX-2 inhibitor treatment | 6 months
  Both left and right fingers were measured twice and the average value was defined as volume of distal part of middle finger
The volume of distal part of middle finger change after COX-2 inhibitor treatment | 12 months
  Both left and right fingers were measured twice and the average value was defined as volume of distal part of middle finger
Circumference of knee joint change after COX-2 inhibitor treatment | 3 months
  During the circumference of knee joint (CKJ) assessment, the patient was standing straight and the knee was extended as much as possible. The tester stood closest to the examined leg and used a tape to measure the circumference just at the base of the patella. Both legs were measured twice and the average value was used as CKJ.
Circumference of knee joint change after COX-2 inhibitor treatment | 6 months
  During the circumference of knee joint (CKJ) assessment, the patient was standing straight and the knee was extended as much as possible. The tester stood closest to the examined leg and used a tape to measure the circumference just at the base of the patella. Both legs were measured twice and the average value was used as CKJ.
Circumference of knee joint change after COX-2 inhibitor treatment | 12 months
  During the circumference of knee joint (CKJ) assessment, the patient was standing straight and the knee was extended as much as possible. The tester stood closest to the examined leg and used a tape to measure the circumference just at the base of the patella. Both legs were measured twice and the average value was used as CKJ.

CONTACTS AND LOCATIONS:
Overall Officials: Weibo Xia, MD, Study Chair — Department of Endocrinology, Key Laboratory of Endocrinology, Ministry of Health, Peking Union Medical College Hospital, Peking Union Medical College, Chinese Academy of Medical Sciences
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China